CLINICAL TRIAL: NCT06799598
Title: DUOSTIM and AI: is There a Difference Between Oocyte Performance in the Follicular and Luteal Phases?
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Yuri Ian Lima Alves de Oliveira, M.D., Rio de Janeiro State University
Other Study IDs: VD001/2025
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DuoStim1: Follicular phase Stimulation
- DuoStim2: Luteal Phase stimulation

SUMMARY:
In vitro fertilization (IVF) has revolutionized assisted reproductive techniques, bringing hope to thousands of people seeking to fulfill their dream of parenthood. However, patients with low ovarian reserve face additional challenges, such as limited response to ovarian stimulation and difficulty in obtaining good-quality eggs. Innovative protocols such as Duostim (dual stimulation) have shown promise in these cases, allowing the maximum number of eggs to be retrieved in a short period of time. In addition, technological advances in the analysis of the quality of mature eggs, such as the use of the Magenta tool, are transforming the way specialists evaluate and select the best gametes to increase the chances of success. This article explores how these approaches complement each other, offering new possibilities for patients with low ovarian reserve and raising the standards of reproductive medicine.

DETAILED DESCRIPTION:
The analysis of the two stimulation phases in a Duostim protocol for IVF using the Magenta tool may have significant clinical relevance, especially in the context of patients with low ovarian reserve or who require optimization in the number of embryos available in IVF cycles in a short period of time. The Magenta tool, being based on AI and machine learning, can identify patterns related to the quality of oocytes and embryos obtained in both phases. This can help determine if there are significant differences in embryo competence between oocytes collected in the follicular phase and the luteal phase. Magenta-powered analysis can provide robust data to validate the Duostim protocol, identify subgroups that benefit most from it, and promote greater clinical efficiency in IVF treatments, especially in challenging cases. This approach can revolutionize the way personalized protocols are designed and monitored to maximize reproductive success. The aim of this study is to compare the two phases of ovarian stimulation - follicular and luteal - in patients undergoing the Duostim protocol, using the Magenta tool for detailed analysis of mature eggs obtained in each phase. The research seeks to identify differences in oocyte quality between the two stages, as well as to evaluate the efficiency of the protocol in maximizing results in patients with low ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF with DUOSTIM protocol and Magenta analysis of mature eggs.

Exclusion Criteria:

* Canceled Duostim Magenta IVF cycles

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women of reproductive age undergoing ovarian stimulation for in vitro fertilization (IVF)
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Follicular and luteal phase oocytes Magenta score | 30 days
  Assessment of oocyte potential to generate blastocysts at two different times of oocyte retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Vida - Medicina Reprodutiva, Rio de Janeiro, Rio de Janeiro, Brazil